CLINICAL TRIAL: NCT04280536
Title: Phase II Study of FTD/TPI (Lonsurf) in Metastatic Breast Cancers With or Without Prior Exposure to Fluoropyrimidines (LONBRECA)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR01/02/19
Record Dates: First submitted 2020-02-10; First posted 2020-02-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: FTD/TPI; TAS-102; Trifluridine
MeSH Terms: conditions — Breast Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: 2 parallel cohorts of patients will be enrolled : Cohort A : patients with prior exposure to fluoropyrimidines Cohort B : patients without prior exposure to fluoropyrimidines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Patients with prior exposure to fluoropyrimidines
  Interventions: Drug: Cohort A
- Cohort B (Experimental): Patients without prior exposure to fluoropyrimidines
  Interventions: Drug: Cohort B

INTERVENTIONS:
Drug: Cohort A — Oral FTD/TPI at RP2D will be administered until disease progression, intolerable toxicity or patient withdrawal.
  Other Names: trifluridine/tipiracil; TAS-102 [Lonsurf]
  Arms: Cohort A
Drug: Cohort B — Oral FTD/TPI at RP2D will be administered until disease progression, intolerable toxicity or patient withdrawal.
  Other Names: trifluridine/tipiracil; TAS-102 [Lonsurf]
  Arms: Cohort B

SUMMARY:
This is a single arm, open-label, lead in phase Ib dose confirmation, followed by phase II study with 2 parallel study cohorts.

DETAILED DESCRIPTION:
Phase Ib Patients will be treated with twice-daily dosing of FTD/TPI in a 3+3 dose escalation design Phase II

Oral FTD/TPI at RP2D will be administered until disease progression, intolerable toxicity or patient withdrawal.

2 parallel cohorts of patients will be enrolled : Cohort A : patients with prior exposure to fluoropyrimidines Cohort B : patients without prior exposure to fluoropyrimidines

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years.
* Histological or cytological diagnosis of breast carcinoma.
* ECOG 0-2.
* HER2 negative tumor (IHC 0 -1+ or IHC 2+ and confirmed on HER2 FISH to be negative based on histological report).
* Patients with HER2 positive tumor may be enrolled if they have failed at least two lines of anti-HER2 based therapies in the metastatic setting, or are intolerant to trastuzumab
* Any hormone receptor status.
* Any number of lines of prior palliative endocrine therapy for patients with hormone receptor positive cancer.
* Has measureable or evaluable disease based on RECIST 1.1 criteria
* Estimated life expectancy of at least 12 weeks.
* Has documented progressive disease from last line of therapy.
* Has recovered from acute toxicities from prior anti-cancer therapies
* Adequate organ function including the following:

oBone marrow: (I) Absolute neutrophil (segmented and bands) count (ANC) ≥1.5 x 109/L (ii) Platelets ≥100 x 109/L (ii) Hemoglobin ≥8 x 109/L oHepatic: (I)Bilirubin ≤ 1.5 x upper limit of normal (ULN), (ii)ALT or AST ≤ 2.5x ULN, (or ≤ 5 X with liver metastases) oRenal: (I) Creatinine ≤1.5x ULN

* Signed informed consent from patient or legal representative.
* Able to comply with study-related procedures.
* Prior therapy (patients enrolled in phase Ib may be enrolled if they fulfil prior therapy criteria for either Cohort A or Cohort B)

  * Cohort A only: Has received at least 2 lines of palliative systemic therapy, including prior fluropyrimidines (capecitabine, TS-1 or 5-fluorouracil) in the palliative setting, or in the adjuvant setting; patients who have only prior exposure to adjuvant fluoropyrimidines must have relapsed within 12 months of completing adjuvant fluoropyrimidines
  * Cohort B only: Any number of prior lines of palliative chemotherapy and has not received fluoropyrimidines (capecitabine, TS-1 or 5-fluorouracil) in the palliative setting or in the adjuvant setting; patients who have prior exposure to adjuvant fluoropyrimidines are eligible if they have relapsed 12 months from completion of adjuvant fluoropyrimidines.

Exclusion Criteria:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Unable to comply with study procedures

Phase Ib lead-in can recruit patients who fulfil criteria for either Cohort A or Cohort B AND all other inclusion/exclusion criteria

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 4 months
  Primary endpoint is proportion of patients who are PFS at 4 months in Cohort A

SECONDARY OUTCOMES:
Overall Response | 5 years
  The death of any patient in the trial from any cause will be recorded and the amount of time from enrollment in the trial until death will be recorded in weeks.
Progression Free Survival (PFS) | 6 months
  Proportion of patients who are PFS at 6 months in Cohort B
Safety and Efficacy | 5 years
  All adverse events experienced by all patients (in both cohort , RP2D of FTD/TPI in MBC Patients) exposed to Trifluridine/tipiracil will be recorded and graded according to CTCAE version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caswell-Jin JL, Plevritis SK, Tian L, Cadham CJ, Xu C, Stout NK, Sledge GW, Mandelblatt JS, Kurian AW. Change in Survival in Metastatic Breast Cancer with Treatment Advances: Meta-Analysis and Systematic Review. JNCI Cancer Spectr. 2018 Nov;2(4):pky062. doi: 10.1093/jncics/pky062. Epub 2018 Dec 24. PMID 30627694
- [Background] Crown J, Dieras V, Kaufmann M, von Minckwitz G, Kaye S, Leonard R, Marty M, Misset JL, Osterwalder B, Piccart M. Chemotherapy for metastatic breast cancer-report of a European expert panel. Lancet Oncol. 2002 Dec;3(12):719-27. doi: 10.1016/s1470-2045(02)00927-0. PMID 12473512